CLINICAL TRIAL: NCT04904211
Title: A National Danish Proof of Concept on Feasiblity and Safety of Home-based Intensive Chemotherapy in Patients With Acute Leukemia.
Brief Title: Feasiblity and Safety of Home-based Intensive Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kristina Holmegaard Nørskov, Clinical Nurse Specialist, PhD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Home-Based Chemo
Record Dates: First submitted 2021-05-22; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Acute Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasiblity and Safety (Experimental): All eligible patients will be assigned to this arm
  Interventions: Other: Home-based chemotherapy

INTERVENTIONS:
Other: Home-based chemotherapy — To investigate the feasibility and safety of home-based intensive chemotherapy in patients with newly diagnosed acute myeloid leukemia (AML) or high-risk myelodysplastic syndrome (MDS). Furthermore, we examined the quality of life (QOL) and psychological wellbeing while receiving induction and consolidation chemotherapy at home.

SUMMARY:
a multicenter single-arm feasibility and safety study of home-based intensive chemotherapy in patients with newly diagnosed acute myeloid leukemia and their quality of life and psychological wellbeing. This national study included patients from six sites in Denmark who received intensive chemotherapy on programmed CADD Solis infusion pumps through a central venous catheter and were also managed as outpatients during treatment-induced pancytopenia.

DETAILED DESCRIPTION:
This national single-arm feasibility cohort study was conducted at six hematology departments at six university hospitals in Denmark: Copenhagen University Hospital, Rigshospitalet; Herlev/Gentofte Hospital; Zealand University Hospital, Roskilde; Odense University Hospital; Aarhus University Hospital, and Aalborg University Hospital.

The project nurse at each site approached and recruited participants from October 2017 to August 2020. The participants were explicitly evaluated for their ability to manage their symptoms, administer oral medication, eat and drink sufficiently, and practice good personal hygiene. Eligible participants received oral and written information and provided written informed consent before inclusion.

Included participants received intensive chemotherapy treatment on a CADD pump through their CVC. The CADD pump is unique because it is portable, carried in a small bag or backpack, and applicable for home-based treatment due to its intuitive and user-friendly interface.

A patient educational program based on strategic patient involvement was integrated into supportive care practice during induction treatment at each hematology department. The program included guidance and training to the patient and/or their primary caregiver in managing the care of their CVC including drawing blood samples, how to use a positive expiratory pressure whistle, functionality of the infusion pump, how to manage and react on pump alarm, and precautions when receiving treatment while being home.

The participants could contact the hematological department from where they received their treatment 24 hours a day by telephone. They were instructed to contact their respective department immediately if fever (>38.0 Celcius) or any pump report alarm occurred. The nurses would then guide the participant to solve the problem from home or recommend they seek help at the department to solve the problem or get evaluated by a doctor.

Adverse events were categorized into non-serious adverse events and serious adverse events. Non-serious adverse events were any pump infusion alarms that could not be solved by phone and required a visit to the hospital. Serious adverse events were any adverse reactions during treatment at home, which resulted in the following outcomes: death or septic shock.

ELIGIBILITY:
Inclusion Criteria:

Participants 18 years or older were included within the first 28 days from diagnosis with AML or high-risk MDS if intensive chemotherapy treatment was planned.

Exclusion Criteria:

Patients were excluded if they did not understand, read and speak Danish, suffered from a severe illness requiring hospitalization if they had an unstable medical disease or any cognitive/psychiatric disorders. During the intervention, participants were withdrawn if hospitalized in an intensive care unit for more than two weeks, if they had a psychological condition (delirium or severe depression), or in case of transition to terminal care or if deceased. Moreover, participants were censored if they relapsed or transitioned to hematopoietic stem cell transplantation (HSCT).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | up to 3 years
  Number of participants included from eligible patients
Adherence to intervention | Up to 24 weeks
  Number of weeks completed out of planned weeks of intervention
Hospital admissions | Up to 24 weeks
  Data will be collected from medical charts
Infections (days) | Up to 24 weeks
  Data will be collected from medical charts
Infections (type) | Up to 24 weeks
  Data will be collected from medical charts
Number of days home during treatment | Up to 24 weeks
  Data will be collected from medical charts
Number of contacts to hospital during treatment | Up to 24 weeks
  Data will be collected from medical charts
Number of removed CVK | Up to 24 weeks
  Data will be collected from medical charts

SECONDARY OUTCOMES:
Psychological wellbeing | Change measures (baseline, 12 weeks, 24 and 36 weeks)
  Measured using the Hospital Anxiety and Depression Scale (HADS)
Quality of Life in participants | Change measures (baseline, 12 weeks, 24 and 36 weeks)
  Measured with the Functional Assessment of Cancer Therapy - Leukemia (FACT-LEU)
Quality of Life in participants | Change measures (baseline, 12 weeks, 24 and 36 weeks)
  Measured with the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30)

CONTACTS AND LOCATIONS:
Locations (6):
- Denmark (6):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense
  - Sjællandsuniversitetshospital Roskilde, Roskilde
  - Rigshospitalet, Copenhagen, Østerbro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Norskov KH, Fridthjof K, Kampmann P, Dunweber A, Andersen CL, Renaberg T, Schollkopf C, Ahmad SA, Schou K, Jensen CF, Moller P, Lundholm BW, Marcher C, Jepsen L, Orntoft AK, Ommen HB, Andersen L, Behrentzs A, Hasselgren CF, Severinsen M, Grand MK, Jarden M, Moller T, Kjeldsen L. A national Danish proof of concept on feasibility and safety of home -based intensive chemotherapy in patients with acute myeloid leukemia. Leuk Res. 2022 Jan;112:106756. doi: 10.1016/j.leukres.2021.106756. Epub 2021 Nov 22. PMID 34839055